CLINICAL TRIAL: NCT04741620
Title: Subacute Effect of Pharmacological Sensory Stimulation of the Oropharynx by Agonists of TRP Receptors in Swallowing Neurophysiology in the Elderly With Oropharyngeal Dysphagia.
Brief Title: Subacute Effect of Pharyngeal Pharmacological Sensory Stimulation in Elderly Patients With Oropharyngeal Dysphagia
Acronym: FIS2018
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Mataró (Other)
Responsible Party: Principal Investigator, Pere Clave, Principal Investigator, Hospital de Mataró
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PI18/00241
Record Dates: First submitted 2021-01-29; First posted 2021-02-05 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Oropharyngeal Dysphagia; Dysphagia; Swallowing Disorder
Keywords: Oropharyngeal dysphagia; TRP agonists; Pharmacological stimulation; Sensory stimulation; Elderly
MeSH Terms: conditions — Deglutition Disorders | interventions — methyl benzoate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Capsaicin 10microM (Active Comparator): 10mL capsaicin 10microM solution 3 times/day during 14 consecutive days (2 weeks).
  Interventions: Other: Piperine 150microM (TRPV1 & TRPA1 natural agonist); Other: Cinnamaldehyde 756,6microM + zinc 70microM (TRPA1 natural agonist); Other: Citric acid 457,5microM (pH=3,5) (ASIC3 natural agonist); Other: Capsaicin 10microM + Citric acid 457,5microM (pH=3,5) (TRPV1 & ASIC3 natural agonists); Other: Placebo (Methyl benzoate, Propyl benzoate, Propylenglycol)
- Piperine 150microM (Active Comparator): 10mL Piperine 150microM solution 3 times/day during 14 consecutive days (2 weeks).
  Interventions: Other: Capsaicin 10microM (TRPV1 natural agonist); Other: Cinnamaldehyde 756,6microM + zinc 70microM (TRPA1 natural agonist); Other: Citric acid 457,5microM (pH=3,5) (ASIC3 natural agonist); Other: Capsaicin 10microM + Citric acid 457,5microM (pH=3,5) (TRPV1 & ASIC3 natural agonists); Other: Placebo (Methyl benzoate, Propyl benzoate, Propylenglycol)
- Cinnamaldehyde 756,6microM + zinc 70microM (Active Comparator): 10mL Cinnamaldehyde 756,6microM + zinc 70microM solution 3 times/day during 14 consecutive days (2 weeks).3 times/day during 14 consecutive days (2 weeks).
  Interventions: Other: Capsaicin 10microM (TRPV1 natural agonist); Other: Piperine 150microM (TRPV1 & TRPA1 natural agonist); Other: Citric acid 457,5microM (pH=3,5) (ASIC3 natural agonist); Other: Capsaicin 10microM + Citric acid 457,5microM (pH=3,5) (TRPV1 & ASIC3 natural agonists); Other: Placebo (Methyl benzoate, Propyl benzoate, Propylenglycol)
- Citric acid 457,5microM (pH=3,5) (Active Comparator): 10mL Citric acid 457,5microM (pH=3,5) solution 3 times/day during 14 consecutive days (2 weeks).3 times/day during 14 consecutive days (2 weeks).
  Interventions: Other: Capsaicin 10microM (TRPV1 natural agonist); Other: Piperine 150microM (TRPV1 & TRPA1 natural agonist); Other: Cinnamaldehyde 756,6microM + zinc 70microM (TRPA1 natural agonist); Other: Capsaicin 10microM + Citric acid 457,5microM (pH=3,5) (TRPV1 & ASIC3 natural agonists); Other: Placebo (Methyl benzoate, Propyl benzoate, Propylenglycol)
- Capsaicin 10microM + Citric acid 457,5microM (pH=3,5) (Active Comparator): 10mL Capsaicin 10microM + Citric acid 457,5microM (pH=3,5) solution 3 times/day during 14 consecutive days (2 weeks).3 times/day during 14 consecutive days (2 weeks).
  Interventions: Other: Capsaicin 10microM (TRPV1 natural agonist); Other: Piperine 150microM (TRPV1 & TRPA1 natural agonist); Other: Cinnamaldehyde 756,6microM + zinc 70microM (TRPA1 natural agonist); Other: Citric acid 457,5microM (pH=3,5) (ASIC3 natural agonist); Other: Placebo (Methyl benzoate, Propyl benzoate, Propylenglycol)
- Placebo (Placebo Comparator): 10mL placebo solution 3 times/day during 14 consecutive days (2 weeks).3 times/day during 14 consecutive days (2 weeks).
  Interventions: Other: Capsaicin 10microM (TRPV1 natural agonist); Other: Piperine 150microM (TRPV1 & TRPA1 natural agonist); Other: Cinnamaldehyde 756,6microM + zinc 70microM (TRPA1 natural agonist); Other: Citric acid 457,5microM (pH=3,5) (ASIC3 natural agonist); Other: Capsaicin 10microM + Citric acid 457,5microM (pH=3,5) (TRPV1 & ASIC3 natural agonists)

INTERVENTIONS:
Other: Capsaicin 10microM (TRPV1 natural agonist) — 10 mL Capsaicin 10microM solution 3 times per day (before each meal) during 14 consecutive days.
  Arms: Capsaicin 10microM + Citric acid 457,5microM (pH=3,5); Cinnamaldehyde 756,6microM + zinc 70microM; Citric acid 457,5microM (pH=3,5); Piperine 150microM; Placebo
Other: Piperine 150microM (TRPV1 & TRPA1 natural agonist) — 10 mL Piperine 150microM solution 3 times per day (before each meal) during 14 consecutive days.
  Arms: Capsaicin 10microM; Capsaicin 10microM + Citric acid 457,5microM (pH=3,5); Cinnamaldehyde 756,6microM + zinc 70microM; Citric acid 457,5microM (pH=3,5); Placebo
Other: Cinnamaldehyde 756,6microM + zinc 70microM (TRPA1 natural agonist) — 10 mL Cinnamaldehyde 756,6microM + zinc 70microM solution 3 times per day (before each meal) during 14 consecutive days.
  Arms: Capsaicin 10microM; Capsaicin 10microM + Citric acid 457,5microM (pH=3,5); Citric acid 457,5microM (pH=3,5); Piperine 150microM; Placebo
Other: Citric acid 457,5microM (pH=3,5) (ASIC3 natural agonist) — 10 mL Citric acid 457,5microM (pH=3,5) solution 3 times per day (before each meal) during 14 consecutive days.
  Arms: Capsaicin 10microM; Capsaicin 10microM + Citric acid 457,5microM (pH=3,5); Cinnamaldehyde 756,6microM + zinc 70microM; Piperine 150microM; Placebo
Other: Capsaicin 10microM + Citric acid 457,5microM (pH=3,5) (TRPV1 & ASIC3 natural agonists) — 10 mL Capsaicin 10microM + Citric acid 457,5microM (pH=3,5) solution 3 times per day (before each meal) during 14 consecutive days.
  Arms: Capsaicin 10microM; Cinnamaldehyde 756,6microM + zinc 70microM; Citric acid 457,5microM (pH=3,5); Piperine 150microM; Placebo
Other: Placebo (Methyl benzoate, Propyl benzoate, Propylenglycol) — 10 mL placebo solution 3 times per day (before each meal) during 14 consecutive days.
  Arms: Capsaicin 10microM; Capsaicin 10microM + Citric acid 457,5microM (pH=3,5); Cinnamaldehyde 756,6microM + zinc 70microM; Citric acid 457,5microM (pH=3,5); Piperine 150microM

SUMMARY:
Oropharyngeal sensory impairments are a potential target for treatment of oropharyngeal dysphagia (OD) in older patients. We previously found acute administration of TRP sensory stimulants improved VFS signs and swallow response. We hypothesized that sub-acute administration of TRP pharyngeal sensory stimulants, would improve cortical neuroplasticity and will lead into a faster and stronger swallow response, however desensitization of TRP receptors may occur. Therefore, the aim of the present study was to assess the biomechanical (Videofluoroscopy) and neurophysiological (pharyngeal sensory evoked potentials -PSEPs- and motor-evoked potentials (MEPs)) effect of 2 week treatment with TRP agonists in older patients with OD. Design: 150 older (>70yr) patients with OD will be included in a Randomized Control Trial assessing the effect of oral administration of either: a) capsaicin (TRPV1); b) piperine (TRPV1/TRPA1) c) cinnamaldehyde (TRPA1); d) citric acid (ASIC3); e) capsaicin+citric acid (TRPV1/ASIC3); and f) placebo (Control). Measurements: 1) VFS signs of safety and efficacy of swallow and timing and extent of swallow response; 2) Latency, amplitude and cortical representation of PSEP and MEP; 3) Substance P concentration in saliva by ELISA as a marker of peripheral stimulation. Results from this study might help to develop new and effective pharmacological treatments for older dysphagic patients, from compensation to recovery of swallow function.

DETAILED DESCRIPTION:
The project consists of a randomized, double-blind controlled interventional clinical trial (patient and analysis of results) with five treatment arms and a control group (placebo) involving a total of 150 elderly patients with oropharyngeal dysphagia (25 patients per group).

The recruitment of participants for the study will be carried out from the patients referred to the Dysphagia Unit of the Hospital de Mataró for the evaluation of swallowing disorders. The swallowing function of all candidates to be included in the study will be clinically evaluated using the volume-viscosity swallowing test (V-VST). Those patients with signs of impaired safety of swallowing during the examination (cough, decreased O2 saturation greater than 2% or voice change) will be candidates to participate in the study. They will be informed and in case of acceptance a saliva sample will be taken, and a videofluoroscopy (VFS) will be performed. If the patient presents impaired safety of swallow (Penetration aspiration scale higher or equal than 2), the patient will be definitively randomized to one of the branches of intervention and the rest of the explorations will proceed (sensory evoked potentials to pharyngeal electrical stimulation and pharyngeal motor evoked potentials to transcranial magnetic stimulation). After the treatment period a second evaluation of study procedures will be performed.

The treatment will consist of administering 10mL solution of the study product, according to randomization, 3 times a day (before breakfast, lunch and dinner) for 14 consecutive days after inclusion in the study. Treatment selected according our previous studies (Alvarez-Berdugo et al. Neurogastroenterol Motil 2017) are: Capsaicin 10microM, Piperine 150microM, Cinnamaldehyde 756,6microM + zinc 70microM, citric acid 457,5microM (pH=3,5), Capsaicin 10microM + citric acid 457,5microM (pH=3,5). For the control group, placebo product will be administered, which will be the vehicle solution with a more neutral pH.

ELIGIBILITY:
Inclusion Criteria:

* More than 70 years old.
* Oropharyngeal dysphagia with impaired safety of swallow (penetration aspiration score higher or equal than 2).
* Patients able to comply with the study protocol.
* Signature or the written informed consent.

Exclusion Criteria:

* Previous history of severe gastrointestinal diseases.
* Epilepsy or previous convulsive crisis episodes.
* Pacemaker or implanted defibrillator carriers.
* Cardiopulmonary instability.
* Oropharyngeal dysphagia of structural cause.
* Previous history of head and neck surgery.
* Neurodegenerative disease.
* Advanced dementia (GDS higher than 5).
* Gastroesophageal reflux.
* Taking drugs with effects on dopamine.
* Neoplasia or active infection.
* Alcohol, tobacco or drugs dependence.
* Participate or have participated in another interventionist clinical trial in the 4 weeks prior to inclusion.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2022-03-27 (Actual); Study Completion 2022-03-27 (Actual)

PRIMARY OUTCOMES:
Change in the score of the Penetration Aspiration Scale | Baseline versus 2/3 days after the intervention
  Differences found in the videofluoroscopy Penetration Aspiration Scale (from 1 (safe swallow) to 8 (silent aspiration)) between treatments and vs. the placebo group.

SECONDARY OUTCOMES:
Impaired safety of swallow | Baseline versus 2/3 days after the intervention
  Videofluoroscopic signs of impaired safety of swallow (penetrations an aspirations)
Impaired efficacy | Baseline versus 2/3 days after the intervention
  Videofluoroscopic signs of impaired efficacy of swallow (oral and pharyngeal residue)
Oropharyngeal swallow response (laryngeal vestibule closure time) | Baseline versus 2/3 days after the intervention
  Laryngeal vestibule closure time (ms) in videofluoroscopy
Oropharyngeal swallow response (upper esophageal opening time) | Baseline versus 2/3 days after the intervention
  Upper esophageal opening time (ms) in videofluoroscopy
Oropharyngeal swallow response (laryngeal vestibule opening time) | Baseline versus 2/3 days after the intervention
  Laryngeal vestibule opening time (ms) in videofluoroscopy
Oropharyngeal swallow response (Bolus final velocity) | Baseline versus 2/3 days after the intervention
  Bolus final velocity (m/s) in videofluoroscopy
Pharyngeal sensory evoked potentials | Baseline versus 2/3 days after the intervention
  Latency and amplitude of N1, P1, N2 and P2 peaks of the Pharyngeal sensory evoked potentials.
Pharyngeal motor evoked potentials | Baseline versus 2/3 days after the intervention
  Latency, amplitude, duration and area under de curve of the Pharyngeal motor evoked potentials.
Sensory threshold | Baseline versus 2/3 days after the intervention
  Sensory threshold to pharyngeal electrical stimulation (mA)
Substance P | Baseline versus 2/3 days after the intervention
  Concentration of substance P in saliva.
Palatability and comfort with the treatment. | Baseline versus 2/3 days after the intervention
  Palatability and comfort with the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Pere Clavé, PhD, Principal Investigator — Hospital de Mataró
Locations (1):
- Consorci Sanitari del Maresme (Hospital de Mataró), Mataró, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guanyabens N, Tomsen N, Palomeras E, Mundet L, Clave P, Ortega O. Neurophysiological characterization of oropharyngeal dysphagia in older patients. Clin Neurophysiol. 2024 Jun;162:129-140. doi: 10.1016/j.clinph.2024.03.030. Epub 2024 Apr 4. PMID 38615499